CLINICAL TRIAL: NCT03524898
Title: NAPAGE: NAb-PAclitaxel and GEmcitabine in Advanced Soft Tissue Sarcoma. A Multicenter Open-label Single Arm Phase Ib/IIa Trial
Brief Title: NAPAGE: NAb-PAclitaxel and GEmcitabine in Advanced Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: As Last patient last visit (LPLV) took place on 15/02/2022, the trial was ended prematurely on this date in accordance with SAKK/CI.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 57/16 - NAPAGE
Record Dates: First submitted 2018-04-24; First posted 2018-05-15 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Soft Tissue Sarcoma
Keywords: Nab-Paclitaxel; Gemcitabine; Advanced soft tissue sarcoma; Cancer; Sarcoma; Abraxane®
MeSH Terms: conditions — Sarcoma; Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: This is a single-arm phase Ib/IIa multi-center study in patients with locally advanced or metastatic soft tissue sarcoma who have received first line or second line chemotherapy with no response or with evidence of disease progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel and gemcitabine (Experimental): Treatment consists of the combination treatment of nab-paclitaxel and gemcitabine, which is given every 2 weeks during 28-day cycle intervals until disease progression.
  Interventions: Drug: Nab-Paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: Nab-Paclitaxel — 150 mg/m2 / 125 mg/m2
  Other Names: Abraxane
Drug: gemcitabine — 1000 mg/m2

SUMMARY:
A clinical trial with biweekly regimen of gemcitabine and nab-paclitaxel for Soft tissue sarcomas (STSs).

A Promising antitumor activity in patients with metastatic STS has been reported with gemcitabine alone or in combination with taxanes including docetaxel and paclitaxel in pre-treated patients.

Nab-paclitaxel is a 130-nm albumin-bound formulation of paclitaxel particles (Celgene, Summit, NJ) which was designed to eliminate the toxicities associated with Cremophor®-EL. Nab-paclitaxel at equal dose of paclitaxel showed increased antitumor activity, enhanced endothelial cell transport and 33% higher intra-tumor paclitaxel concentration in preclinical models of solid tumor xenografts promising an advantageous pharmacokinetic profile In sarcoma, nab-paclitaxel demonstrated preclinical anti-tumor activity in rhabdomyosarcoma xenograft model. Local relapsed tumors following paclitaxel treatment proved to be paclitaxel-resistant but remained responsive to nab-paclitaxel.

These findings provide the rationale for further evaluation of nab-paclitaxel in combination with gemcitabine for soft tissue sarcoma treatment.

DETAILED DESCRIPTION:
Soft tissue sarcomas (STSs) account for 1% of all human cancers and consist of at least 50 different histological subtypes which have different clinical behavior and response to chemotherapy. Patients with advanced disease (locally advanced or metastatic) have a somber prognosis with a median OS between 12 and 15 months.

Palliative chemotherapy is the mainstay of treatment in the metastatic setting, although in a small subset with limited metastases local treatment may be curative. First-line treatment for advanced soft-tissue sarcoma includes doxorubicin hydrochloride, alone or in combination with other chemotherapy agents (e.g., ifosfamide), or olaratumab. Beyond first line several agents have shown activity, including gemcitabine/docetaxel, trabectedin and pazopanib, though no standard regimen has been established.

Promising antitumor activity in patients with metastatic STS has been reported with gemcitabine alone or in combination with taxanes including docetaxel and paclitaxel in pre-treated patients.

Nab-paclitaxel is a 130-nm albumin-bound formulation of paclitaxel particles (Abraxane®, Celgene, Summit, NJ) which was designed to eliminate the toxicities associated with Cremophor EL®. Nab-paclitaxel at equal dose of paclitaxel showed increased antitumor activity, enhanced endothelial cell transport and 33% higher intra-tumor paclitaxel concentration in preclinical models of solid tumor xenografts promising an advantageous pharmacokinetic profile In sarcoma, nab-paclitaxel demonstrated preclinical antitumor activity in rhabdomyosarcoma xenograft model. Local relapsed tumors following paclitaxel treatment proved to be paclitaxel-resistant but remained responsive to nab-paclitaxel.

These findings provide the rationale for further evaluation of nab-paclitaxel in combination with gemcitabine for soft tissue sarcoma treatment.

Phase Ib objective:

* To assess the safety and feasibility of combining nab-paclitaxel and gemcitabine

Phase II objective:

* To determine whether or not gemcitabine/nab-paclitaxel regimen exhibits antitumor activity that is worth testing further in STS.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed minimum grade 2, locally advanced or metastatic STS refractory to chemotherapy and not suitable for local treatment.
* Minimum one line and maximum 2 lines of previous chemotherapy for advanced/metastatic STS
* Measurable disease according to RECIST v1.1
* Age ≥ 18 years
* WHO performance status 0-2
* Adequate hematological, hepatic and renal function
* Negative pregnancy test
* Effective method of birth control
* Peripheral neuropathy at enrolment must be ≤ grade 1

Exclusion Criteria:

* Uncontrolled CNS metastases
* Previous or concomitant malignancy diagnosed within 3 years
* More than 2 lines of previous systemic treatment for STS
* Previous sarcoma treatment with gemcitabine and/or nab-paclitaxel or other taxanes
* Radiotherapy within 4 weeks prior to registration
* Concurrent or recent treatment with any other experimental drug
* Concomitant use of other anti-cancer drugs
* Severe or uncontrolled cardiovascular disease
* History of cerebrovascular accident or intracranial hemorrhage within 2 months prior to registration
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information
* Known hypersensitivity to the trial drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose-limiting toxicity (DLT) | during the first cycle of treatment (28 days)
  DLT is defined as any of the following adverse events (AEs) occurring during the first cycle of treatment and regarded by the investigators and/or the Sponsor to be related to nab-paclitaxel and/or gemcitabine (AEs not related to the IMPs are not regarded as DLT)
Phase II: Progression-free rate (PFR) | at 12 weeks after registration
  PFR at 12 weeks after registration determined by the percentage of progression-free patients at 12 weeks. Progression is defined as one of the following events (whichever occurs first):
  * Progressive disease (PD) assessed according to the RECIST v1.1 before week 13 (allowed is a 1 week delay in the tumor assessment at week 12).
  * Death due to any cause up to week 12.
  * Start of second line treatment before week 12.
  * No tumor assessment after week 11 without subsequent treatment which shows stabilization or response.

SECONDARY OUTCOMES:
Phase I: PFR 12 weeks | at 12 weeks after registration
Phase I: Best response assessed according to RECIST v1.1 | assessed for up to 5 years after patient registration
Phase I: Adverse events (AEs), assessed according to NCI CTCAE v4.03 | assessed for up to 5 years after patient registration
Phase II: Progression-free survival (PFS) | assessed for up to 5 years after patient registration
  PFS defined as the time from registration until progression according to RECIST v1.1 or death from any cause, whichever occurs first.
  Patients without an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of the last tumor assessment before the start of the new therapy, if any.
Phase II: Overall Survival (OS) | assessed for up to 5 years after patient registration
  OS defined as the time from registration until death from any cause. Patients without an event at the time of analysis will be censored at the date they were last known to be alive.
Phase II: Best response assessed according to RECIST v1.1 | assessed for up to 5 years after patient registration
Phase II: AEs, assessed according to NCI CTCAE v4.03 | from registration until 28 days after administration of the last dose of trial treatment
Phase II: Symptom-related quality of life assessed by questionnaires | assessed for up to 5 years after patient registration
  Symptom-related quality of life will be assessed with the M.D. Anderson Symptom Inventory (MDASI), which measures the severity of 13 cancer-related symptoms and their impact on six dimensions of daily life at their worst in the last 24 hours on a 0-10 numerical rating scale, with 0 being "not present" and 10 being "as bad as you can imagine."
Phase II: Nab-paclitaxel related sensory neuropathy assessed by questionnaires | assessed for up to 5 years after patient registration
  To address an important side-effect of nab-paclitaxel, sensory neuropathy will be assessed by the 4-item subscale of the FACT/GOG-Ntx (Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity), which measures the severity of sensory neuropathy in the last 7 days on a 0-4 numerical rating scale, with 0 being "not at all" and 4 being "very much."

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Digklia, MD, Study Chair — Département d'Oncologie CHUV , Lausanne; Christian Rothermundt, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (8):
- Switzerland (8):
  - Universitaetsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital, Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - CHUV - Swiss Cancer Center Lausanne, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No